CLINICAL TRIAL: NCT02563353
Title: PTH and Vibration in OSteoporosis (PaVOS) Study
Brief Title: PTH and Vibration in OSteoporosis Study
Acronym: PaVOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Copenhagen University Hospital, Denmark (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Sygehus Lillebaelt (Other); Odense Patient Data Explorative Network (Other); Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Lars Matzen, MD, Clin. Ass. Professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20150121
Record Dates: First submitted 2015-09-15; First posted 2015-09-30 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Osteoporosis
Keywords: whole body vibration; PTH
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- controlgroup (Active Comparator): Teriparatide, 20 microgram/day. 24 months of treatment
  Interventions: Drug: teriparatide
- studygroup 1 (Experimental): Teriparatide, 20 microgram/day. 24 months of treatment.
  12 months of Whole-body vibration on vibration platforms.
  Interventions: Other: whole-body vibration; Drug: teriparatide
- studygroup 2 (Experimental): Teriparatide, 20 microgram/day. 24 months of treatment.
  24 months of Whole-body vibration on vibration platforms
  Interventions: Other: whole-body vibration; Drug: teriparatide

INTERVENTIONS:
Other: whole-body vibration — Whole-body vibration on vibration platforms. 30-40 Hertz, from 2 mm (low) to 4 mm (high) amplitude,
  1 minutes x 6 with 1 minute break between. 3 times a week.
  Other Names: vibration therapy
  Arms: studygroup 1; studygroup 2
Drug: teriparatide — Teriparatide, 20 microgram/day. 24 months of treatment.
  Other Names: PTH

SUMMARY:
Objective:

This is a randomized controlled trial (RCT) in osteoporosis patients randomized to standard parathyroid hormone (PTH) treatment alone or to standard PTH treatment and Whole-body vibration (WBV). PTH is an effective but expensive anabolic treatment for osteoporosis. WBV stimulates muscles and bones. A combined treatment might have synergistic or additive beneficial effects on bone, reducing fracture risk making treatment more effective and cost-effective. A beneficial effect on muscles and thereby falls risk of WBV may improve fracture risk even further.

If the results of this pilot study are promising then a strong case can be made for a large multi-centre RCT using strong endpoints including fractures and falls.

DETAILED DESCRIPTION:
Study Objectives

1. To determine if WBV in addition to standard PTH treatment has a greater effect on bone mass in osteoporosis patients compared to standard PTH treatment alone.
2. To determine if WBV in addition to standard PTH treatment has a greater effect on bone microarchitecture in osteoporosis patients compared to standard PTH treatment alone, as assessed by high resolution peripheral quantitative computed tomography (HR-pQCT).
3. To determine if WBV in addition to standard PTH treatment has a greater effect on markers of bone formation and resorption in osteoporosis patients compared to standard PTH treatment alone.
4. To study the effects of WBV on muscle function and balance in osteoporosis
5. To assess the safety and adherence to WBV in osteoporotic patients

Study Design:

General Design This will be a multi-center randomized controlled trial (RCT) in osteoporosis patients being started on standard PTH treatment according to Danish Osteoporosis guidelines. Participants will be randomized to standard PTH treatment alone or to standard PTH treatment and WBV.

Statistical Plan:

Sample Size Determination The inclusion of 32 participants (16 in both groups) would give the study 80% power to detect a clinically significant additional increase of 22% with WBV (assuming a 9% increase of BMD in the PTH alone group and 11% increase in the combined PTH+WBV group, and assuming a SD of the BMD increase of 2%. Allowing for a 20% dropout rate, the plan is to include 40 participants (20 in each group). From previous research on WBV by one of the investigators (TM), statistically significant differences were found in bone formation markers and in muscle strength at 3 months between the WBV and control groups with a sample size of 35. The number of participants in the latter pilot work is reassuringly consistent with the sample size calculations. The number needed to be included is far less (34%) than the actual number of patients treated with PTH in the recruiting departments in a similar time period last year.

Statistical Methods:

STATA/SPSS will be used for data analysis. For the primary endpoint (BMD at 12 months) the mean percentage changes in BMD between the two groups will be compared using Analysis of Variance (ANOVA) provided the distribution is normal. For the other endpoints parametric tests will be used to assess differences in the two groups for normally distributed data and non-parametric tests for data not normally distributed.

The randomization will be done online in the data capture program Red Cap. There will be created a Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, and normal ranges if relevant.

Information:

Participants will be recruited during their attendance at the outpatient clinics. At that time the subjects will be given a full explanation of the study as well as the patient information sheet and invited to participate in the study. At an interval of not less than 24 hours, patients will be invited to consent prior to starting their PTH treatment.

The information will be sufficient for subjects to make an informed decision about their participation in this study. The subject will complete and sign a consent form to indicate they are giving valid consent to participate in the trial.

Withdrawal of Subjects:

Patients who withdraw consent from participation in the trial will be withdrawn from the trial. This will not affect their standard medical management and not cause any adverse effect on the subject.

ELIGIBILITY:
Inclusion Criteria:

* Women starting PTH treatment for osteoporosis according to Danish Osteoporosis guidelines

Exclusion Criteria:

* Women currently taking oral glucocorticoids
* Women unable to give informed consent
* Women unable to stand for 2 minutes at a time on the vibration platform
* Women who have contraindications to WBV (e.g. joint prosthesis, pacemakers)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Changes in the BMD, Bone Mineral Density of hip and spine region (Hologic DXA machine) | at the time the participants start treatment and in an interval as close as possible to after 6, 12, 18, 24 months from baseline
  DXA scan of hip and spine regions, BMD (g/cm^2)

SECONDARY OUTCOMES:
Changes in the Bone microarchitecture at the tibia | at the time the participants start treatment and in an interval as close as possible to after 6, 12, 18 and 24 months from baseline
  HRpQCT assesses parameters of bone microarchitecture at the tibia.
Changes in the Bone microarchitecture at the radius | at the time the participants start treatment and in an interval as close as possible to after 6, 12, 18 and 24 months from baseline
  HRpQCT assesses parameters of bone microarchitecture at the radius.
changes in muscle mass | at the time the participants start treatment and in an interval as close as possible to after 12 and 24 months from baseline
  Full body DXA
Changes from baseline in the markers of bone resorption | at the time the participants start treatment and in an interval as close as possible to after 3, 6, 12, 18, 24 months from baseline
  CTX, sclerostin
Changes from baseline in the markers of bone formation | at the time the participants start treatment and in an interval as close as possible to after 3, 6, 12, 18, 24 months from baseline
  P1NP
Changes in Muscle strength | at the time the participants start treatment and in an interval as close as possible to after 3,6,12,18 and 24 months from baseline
  Measurements of muscle strength (leg extensor power)
Changes in handgrip strength | at the time the participants start treatment and in an interval as close as possible to after 3,6,12,18 and 24 months from baseline
  Measurements of muscle strength (handgrip strength)
Changes in Balance | at the time the participants start treatment and in an interval as close as possible to after 3, 6 ,12, 18 and 24 months from baseline
  Short Physical Performance Battery (SPPB)
Adherence to WBV | During 2 years from the start of the treatment
  Self Reporting training log
Changes in physical activity | at the time the participants start treatment and in an interval as close as possible to after 12, and 24 months from baseline
  IPAQ short version
Changes in quality of life | at the time the participants start treatment and in an interval as close as possible to after 12, and 24 months from baseline
  EQ5D questionaire.
Changes in basic mobility | at the time the participants start treatment and in an interval as close as possible to after 3,6,12,18 and 24 months from baseline
  Time up and go test
Changes in The Falls Efficacy Scale International | at the time the participants start treatment and in an interval as close as possible to after 12, and 24 months from baseline
  FES-I

CONTACTS AND LOCATIONS:
Overall Officials: Lars Matzen, Clin.Ass.Pro, Principal Investigator — Odense University Hospital; Ditte Jepsen, MD, ph.d. student, Principal Investigator — University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] O'Neill TW, Cockerill W, Matthis C, Raspe HH, Lunt M, Cooper C, Banzer D, Cannata JB, Naves M, Felsch B, Felsenberg D, Janott J, Johnell O, Kanis JA, Kragl G, Lopes Vaz A, Lyritis G, Masaryk P, Poor G, Reid DM, Reisinger W, Scheidt-Nave C, Stepan JJ, Todd CJ, Woolf AD, Reeve J, Silman AJ. Back pain, disability, and radiographic vertebral fracture in European women: a prospective study. Osteoporos Int. 2004 Sep;15(9):760-5. doi: 10.1007/s00198-004-1615-4. Epub 2004 May 12. PMID 15138664
- [Background] Cockerill W, Lunt M, Silman AJ, Cooper C, Lips P, Bhalla AK, Cannata JB, Eastell R, Felsenberg D, Gennari C, Johnell O, Kanis JA, Kiss C, Masaryk P, Naves M, Poor G, Raspe H, Reid DM, Reeve J, Stepan J, Todd C, Woolf AD, O'Neill TW. Health-related quality of life and radiographic vertebral fracture. Osteoporos Int. 2004 Feb;15(2):113-9. doi: 10.1007/s00198-003-1547-4. Epub 2003 Nov 13. PMID 14618303
- [Background] Tosteson AN, Gabriel SE, Grove MR, Moncur MM, Kneeland TS, Melton LJ 3rd. Impact of hip and vertebral fractures on quality-adjusted life years. Osteoporos Int. 2001 Dec;12(12):1042-9. doi: 10.1007/s001980170015. PMID 11846331
- [Background] Borgstrom F, Zethraeus N, Johnell O, Lidgren L, Ponzer S, Svensson O, Abdon P, Ornstein E, Lunsjo K, Thorngren KG, Sernbo I, Rehnberg C, Jonsson B. Costs and quality of life associated with osteoporosis-related fractures in Sweden. Osteoporos Int. 2006;17(5):637-50. doi: 10.1007/s00198-005-0015-8. Epub 2005 Nov 9. PMID 16283064
- [Background] Burge R, Dawson-Hughes B, Solomon DH, Wong JB, King A, Tosteson A. Incidence and economic burden of osteoporosis-related fractures in the United States, 2005-2025. J Bone Miner Res. 2007 Mar;22(3):465-75. doi: 10.1359/jbmr.061113. PMID 17144789
- [Background] Neer RM, Arnaud CD, Zanchetta JR, Prince R, Gaich GA, Reginster JY, Hodsman AB, Eriksen EF, Ish-Shalom S, Genant HK, Wang O, Mitlak BH. Effect of parathyroid hormone (1-34) on fractures and bone mineral density in postmenopausal women with osteoporosis. N Engl J Med. 2001 May 10;344(19):1434-41. doi: 10.1056/NEJM200105103441904. PMID 11346808
- [Background] Blick SK, Dhillon S, Keam SJ. Teriparatide: a review of its use in osteoporosis. Drugs. 2008;68(18):2709-37. doi: 10.2165/0003495-200868180-00012. PMID 19093708
- [Background] Bergmann P, Body JJ, Boonen S, Boutsen Y, Devogelaer JP, Goemaere S, Kaufman J, Reginster JY, Rozenberg S. Loading and skeletal development and maintenance. J Osteoporos. 2010 Dec 20;2011:786752. doi: 10.4061/2011/786752. PMID 21209784
- [Background] Lewis RD, Modlesky CM. Nutrition, physical activity, and bone health in women. Int J Sport Nutr. 1998 Sep;8(3):250-84. doi: 10.1123/ijsn.8.3.250. PMID 9738135
- [Background] Rizzoli R, Bianchi ML, Garabedian M, McKay HA, Moreno LA. Maximizing bone mineral mass gain during growth for the prevention of fractures in the adolescents and the elderly. Bone. 2010 Feb;46(2):294-305. doi: 10.1016/j.bone.2009.10.005. Epub 2009 Oct 17. PMID 19840876
- [Background] Chow JW, Fox S, Jagger CJ, Chambers TJ. Role for parathyroid hormone in mechanical responsiveness of rat bone. Am J Physiol. 1998 Jan;274(1):E146-54. doi: 10.1152/ajpendo.1998.274.1.E146. PMID 9458760
- [Background] Li J, Duncan RL, Burr DB, Gattone VH, Turner CH. Parathyroid hormone enhances mechanically induced bone formation, possibly involving L-type voltage-sensitive calcium channels. Endocrinology. 2003 Apr;144(4):1226-33. doi: 10.1210/en.2002-220821. PMID 12639904
- [Background] Roberts MD, Santner TJ, Hart RT. Local bone formation due to combined mechanical loading and intermittent hPTH-(1-34) treatment and its correlation to mechanical signal distributions. J Biomech. 2009 Nov 13;42(15):2431-8. doi: 10.1016/j.jbiomech.2009.08.030. Epub 2009 Sep 26. PMID 19782988
- [Background] Wysocki A, Butler M, Shamliyan T, Kane RL. Whole-body vibration therapy for osteoporosis: state of the science. Ann Intern Med. 2011 Nov 15;155(10):680-6, W206-13. doi: 10.7326/0003-4819-155-10-201111150-00006. PMID 22084334
- [Background] Gusi N, Raimundo A, Leal A. Low-frequency vibratory exercise reduces the risk of bone fracture more than walking: a randomized controlled trial. BMC Musculoskelet Disord. 2006 Nov 30;7:92. doi: 10.1186/1471-2474-7-92. PMID 17137514
- [Background] Cardinale M, Pope MH. The effects of whole body vibration on humans: dangerous or advantageous? Acta Physiol Hung. 2003;90(3):195-206. doi: 10.1556/APhysiol.90.2003.3.2. PMID 14594190
- [Background] Cardinale M, Rittweger J. Vibration exercise makes your muscles and bones stronger: fact or fiction? J Br Menopause Soc. 2006 Mar;12(1):12-8. doi: 10.1258/136218006775997261. PMID 16513017
- [Background] Cardinale M, Wakeling J. Whole body vibration exercise: are vibrations good for you? Br J Sports Med. 2005 Sep;39(9):585-9; discussion 589. doi: 10.1136/bjsm.2005.016857. PMID 16118292
- [Background] Eisman JA. Good, good, good... good vibrations: the best option for better bones? Lancet. 2001 Dec 8;358(9297):1924-5. doi: 10.1016/S0140-6736(01)06975-6. No abstract available. PMID 11747912
- [Background] Rubin C, Xu G, Judex S. The anabolic activity of bone tissue, suppressed by disuse, is normalized by brief exposure to extremely low-magnitude mechanical stimuli. FASEB J. 2001 Oct;15(12):2225-9. doi: 10.1096/fj.01-0166com. PMID 11641249
- [Background] Xie L, Jacobson JM, Choi ES, Busa B, Donahue LR, Miller LM, Rubin CT, Judex S. Low-level mechanical vibrations can influence bone resorption and bone formation in the growing skeleton. Bone. 2006 Nov;39(5):1059-1066. doi: 10.1016/j.bone.2006.05.012. Epub 2006 Jul 7. PMID 16824816
- [Background] Judex S, Lei X, Han D, Rubin C. Low-magnitude mechanical signals that stimulate bone formation in the ovariectomized rat are dependent on the applied frequency but not on the strain magnitude. J Biomech. 2007;40(6):1333-9. doi: 10.1016/j.jbiomech.2006.05.014. Epub 2006 Jun 30. PMID 16814792
- [Background] Xie L, Rubin C, Judex S. Enhancement of the adolescent murine musculoskeletal system using low-level mechanical vibrations. J Appl Physiol (1985). 2008 Apr;104(4):1056-62. doi: 10.1152/japplphysiol.00764.2007. Epub 2008 Feb 7. PMID 18258802
- [Background] Rubin C, Pope M, Fritton JC, Magnusson M, Hansson T, McLeod K. Transmissibility of 15-hertz to 35-hertz vibrations to the human hip and lumbar spine: determining the physiologic feasibility of delivering low-level anabolic mechanical stimuli to skeletal regions at greatest risk of fracture because of osteoporosis. Spine (Phila Pa 1976). 2003 Dec 1;28(23):2621-7. doi: 10.1097/01.BRS.0000102682.61791.C9. PMID 14652479
- [Background] Bosco C, Iacovelli M, Tsarpela O, Cardinale M, Bonifazi M, Tihanyi J, Viru M, De Lorenzo A, Viru A. Hormonal responses to whole-body vibration in men. Eur J Appl Physiol. 2000 Apr;81(6):449-54. doi: 10.1007/s004210050067. PMID 10774867
- [Background] Erskine J, Smillie I, Leiper J, Ball D, Cardinale M. Neuromuscular and hormonal responses to a single session of whole body vibration exercise in healthy young men. Clin Physiol Funct Imaging. 2007 Jul;27(4):242-8. doi: 10.1111/j.1475-097X.2007.00745.x. PMID 17564674
- [Background] Fritton JC, Rubin CT, Qin YX, McLeod KJ. Whole-body vibration in the skeleton: development of a resonance-based testing device. Ann Biomed Eng. 1997 Sep-Oct;25(5):831-9. doi: 10.1007/BF02684167. PMID 9300107
- [Background] Gilsanz V, Wren TA, Sanchez M, Dorey F, Judex S, Rubin C. Low-level, high-frequency mechanical signals enhance musculoskeletal development of young women with low BMD. J Bone Miner Res. 2006 Sep;21(9):1464-74. doi: 10.1359/jbmr.060612. PMID 16939405
- [Background] Cardinale M, Lim J. Electromyography activity of vastus lateralis muscle during whole-body vibrations of different frequencies. J Strength Cond Res. 2003 Aug;17(3):621-4. doi: 10.1519/1533-4287(2003)0172.0.co;2. PMID 12930196
- [Background] Hazell TJ, Kenno KA, Jakobi JM. Evaluation of muscle activity for loaded and unloaded dynamic squats during vertical whole-body vibration. J Strength Cond Res. 2010 Jul;24(7):1860-5. doi: 10.1519/JSC.0b013e3181ddf6c8. PMID 20543737
- [Background] Roelants M, Verschueren SM, Delecluse C, Levin O, Stijnen V. Whole-body-vibration-induced increase in leg muscle activity during different squat exercises. J Strength Cond Res. 2006 Feb;20(1):124-9. doi: 10.1519/R-16674.1. PMID 16503671
- [Background] Pollock RD, Woledge RC, Mills KR, Martin FC, Newham DJ. Muscle activity and acceleration during whole body vibration: effect of frequency and amplitude. Clin Biomech (Bristol). 2010 Oct;25(8):840-6. doi: 10.1016/j.clinbiomech.2010.05.004. Epub 2010 Jun 11. PMID 20541297
- [Background] Russo CR, Lauretani F, Bandinelli S, Bartali B, Cavazzini C, Guralnik JM, Ferrucci L. High-frequency vibration training increases muscle power in postmenopausal women. Arch Phys Med Rehabil. 2003 Dec;84(12):1854-7. doi: 10.1016/s0003-9993(03)00357-5. PMID 14669194
- [Background] Torvinen S, Kannu P, Sievanen H, Jarvinen TA, Pasanen M, Kontulainen S, Jarvinen TL, Jarvinen M, Oja P, Vuori I. Effect of a vibration exposure on muscular performance and body balance. Randomized cross-over study. Clin Physiol Funct Imaging. 2002 Mar;22(2):145-52. doi: 10.1046/j.1365-2281.2002.00410.x. PMID 12005157
- [Background] Ward K, Alsop C, Caulton J, Rubin C, Adams J, Mughal Z. Low magnitude mechanical loading is osteogenic in children with disabling conditions. J Bone Miner Res. 2004 Mar;19(3):360-9. doi: 10.1359/JBMR.040129. Epub 2004 Jan 27. PMID 15040823
- [Background] Tanaka SM, Alam IM, Turner CH. Stochastic resonance in osteogenic response to mechanical loading. FASEB J. 2003 Feb;17(2):313-4. doi: 10.1096/fj.02-0561fje. Epub 2002 Dec 3. PMID 12475888
- [Background] Kerschan-Schindl K, Grampp S, Henk C, Resch H, Preisinger E, Fialka-Moser V, Imhof H. Whole-body vibration exercise leads to alterations in muscle blood volume. Clin Physiol. 2001 May;21(3):377-82. doi: 10.1046/j.1365-2281.2001.00335.x. PMID 11380538
- [Background] Corrie H, Brooke-Wavell K, Mansfield NJ, Cowley A, Morris R, Masud T. Effects of vertical and side-alternating vibration training on fall risk factors and bone turnover in older people at risk of falls. Age Ageing. 2015 Jan;44(1):115-22. doi: 10.1093/ageing/afu136. Epub 2014 Oct 7. PMID 25294839
- [Background] Verschueren SM, Roelants M, Delecluse C, Swinnen S, Vanderschueren D, Boonen S. Effect of 6-month whole body vibration training on hip density, muscle strength, and postural control in postmenopausal women: a randomized controlled pilot study. J Bone Miner Res. 2004 Mar;19(3):352-9. doi: 10.1359/JBMR.0301245. Epub 2003 Dec 22. PMID 15040822
- [Background] Gomez-Cabello A, Ara I, Gonzalez-Aguero A, Casajus JA, Vicente-Rodriguez G. Effects of training on bone mass in older adults: a systematic review. Sports Med. 2012 Apr 1;42(4):301-25. doi: 10.2165/11597670-000000000-00000. PMID 22376192
- [Background] Sitja Rabert M, Rigau Comas D, Fort Vanmeerhaeghe A, Santoyo Medina C, Roque i Figuls M, Romero-Rodriguez D, Bonfill Cosp X. Whole-body vibration training for patients with neurodegenerative disease. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD009097. doi: 10.1002/14651858.CD009097.pub2. PMID 22336858
- [Derived] Jepsen DB, Masud T, Holsgaard-Larsen A, Hansen S, Jorgensen NR, Ryg J. The combined effect of parathyroid hormone (1-34) and whole-body vibration exercise on physical performance in OSteoporotic women (PaVOS study): a secondary analysis from a randomised controlled trial. BMC Sports Sci Med Rehabil. 2020 Sep 5;12:54. doi: 10.1186/s13102-020-00204-w. eCollection 2020. PMID 32944251
- [Derived] Jepsen DB, Ryg J, Hansen S, Jorgensen NR, Gram J, Masud T. The combined effect of Parathyroid hormone (1-34) and whole-body Vibration exercise in the treatment of postmenopausal OSteoporosis (PaVOS study): a randomized controlled trial. Osteoporos Int. 2019 Sep;30(9):1827-1836. doi: 10.1007/s00198-019-05029-z. Epub 2019 Jul 15. PMID 31309239
- [Derived] Jepsen DB, Ryg J, Jorgensen NR, Hansen S, Masud T. The combined effect of Parathyroid hormone (1-34) and whole-body Vibration exercise in the treatment of OSteoporosis (PaVOS)- study protocol for a randomized controlled trial. Trials. 2018 Mar 16;19(1):186. doi: 10.1186/s13063-018-2551-5. PMID 29548300